CLINICAL TRIAL: NCT04071028
Title: Heart Rate Variability as an Indicator Associated With the Improvement of Dysmenorrhea After the Warm-water Footbath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camillians Saint Mary's Hospital Luodong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMHL_HRVnFB
Record Dates: First submitted 2019-08-06; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Primary Dysmenorrhea
Keywords: footbath; parasympathetic activity; primary dysmenorrhea; sympathetic activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Footbath group (Active Comparator): All the participants were arranged to stay in an air-conditioned, quiet room from 5:30 to 6:30 p.m. on their menstruation days 1 and 2. After sitting quietly for 20 minutes, the participants in the "footbath group" received legs soaking from the heel to the Sanyinjiao (SP6) acupoint (above the ankle) 24 in 42 ℃ water with air bubbles and vibration given to the soles for 20 minutes,
  Interventions: Procedure: warm-water footbath
- Control group (No Intervention): All the participants were arranged to stay in an air-conditioned, quiet room from 5:30 to 6:30 p.m. on their menstruation days 1 and 2. After sitting quietly for 20 minutes, whereas the participants in the "control group" kept on sitting quietly without legs soaking during the additional 20-minute period.

INTERVENTIONS:
Procedure: warm-water footbath — All the participants in the intervention group were arranged to stay in an air-conditioned, quiet room from 5:30 to 6:30 p.m. on their menstruation days 1 and 2. After sitting quietly for 20 minutes, the participants in the "footbath group" received legs soaking from the heel to the Sanyinjiao (SP6) acupoint (above the ankle) 24 in 42 ℃ water with air bubbles and vibration given to the soles for 20 minutes, whereas the participants in the "control group" kept on sitting quietly without legs soaking during the additional 20-minute period.
  Arms: Footbath group

SUMMARY:
The effect of warm-water footbath in improving primary dysmenorrhea (PD) was rarely investigated previously. We aimed to exam the hypothesis that warm-water footbath is effective to reduce the pain of PD, and the effect is associated with changes in the autonomic nervous system (ANS) activity.

The quasi-experimental study was carried out enrolling 68 college students) with PD. The enrolled participants were randomized into two groups and received interventions (footbath (n=35) versus sitting only (n=33)) for 20 minutes per day on their menstruation days 1 and 2.

After the interventions, we analyzed the association among intervention (with footbath versus without footbath), heart rate variability (HRV) changes and changes of pain scales (Pain Visual Analog Scale and short-form McGill Pain Questionnaire).

DETAILED DESCRIPTION:
Dysmenorrhea is the most common gynecological condition affecting 16% to 95% of adolescents and young women, and reduce their quality of life. Primary dysmenorrhea (PD), a term denoting the dysmenorrhea in the absence of underlying pathology, is commonly referred to as period pain or menstrual cramps by the lay press and public.

The effect of warm-water footbath in improving primary dysmenorrhea (PD) was rarely investigated previously. We aimed to exam the hypothesis that warm-water footbath is effective to reduce the pain of PD, and the effect is associated with changes in the autonomic nervous system (ANS) activity.

This study was approved by the Institutional Review Board of Saint Mary Hospital Luodong (SMHIRB102015).

This study with a quasi-experimental design was conducted in a nursing college in Northern Taiwan during the study period from December 1, 2013, to June 30, 2014. Participants were eligible for enrollment if they: (1) were healthy female students aged 16-20 years of the nursing college; (2) had regular menstrual cycles; (3) experienced dysmenorrhea within 6 months before the enrollment; (4) had dysmenorrhea with severity higher than five scores of the pain visual analog scale (PVAS); and (5) had no experience of pregnancy. The exclusion criteria included individuals whom: (1) had irregular menstrual cycles; (2) had circulation problem of legs such as peripheral arterial occlusive disease or deep vein thrombosis; (3) had wounds or skin lesions over legs; and (4) had taken any medications which affect ANS activity. The suggested participant's number estimated by the G-Power was 34 when setting the calculated power as 0.8 and α as 0.05. Considering participant loss during the study process, we decided to enroll 68 participants.

All enrolled participants were randomized into the footbath group (n=35) and control group (n=33). The baseline demographic data, as well as relevant information about menstrual cycles and dysmenorrhea of all participants, were documented at enrollment. All the participants were arranged to stay in an air-conditioned, quiet room from 5:30 to 6:30 p.m. on their menstruation days 1 and 2. After sitting quietly for 20 minutes, the participants in the "footbath group" received legs soaking from the heel to the Sanyinjiao (SP6) acupoint (above the ankle) 24 in 42 ℃ water with air bubbles and vibration given to the soles for 20 minutes, whereas the participants in the "control group" kept on sitting quietly without legs soaking during the additional 20-minute period.

PVAS and Short-Form McGill Pain Questionnaire (SF-MPQ) were fulfilled as pain assessment by all participants twice, including a "pre-test" before the intervention of menstruation day 1 and a "post-test" after the intervention of menstruation day 2.

HRV was measured at four time points (before and immediately after the interventions on days 1 and 2) to assess ANS function for all participants.

The interventions were "warm-water footbath for 20 minutes" for the "footbath group" and "sitting quietly without footbath for 20 minutes" for the "control group." Then we evaluated the influence of warm-water footbath on dysmenorrhea and several variables, including HRV indices and stiffness index.

ELIGIBILITY:
Inclusion criteria:

1. healthy female students aged 16-20 years of the nursing college;
2. had regular menstrual cycles;
3. experienced dysmenorrhea within 6 months before the enrollment;
4. had dysmenorrhea with severity higher than five scores of the pain visual analog scale (PVAS); and
5. had no experience of pregnancy.

Exclusion criteria:

1. had irregular menstrual cycles;
2. had circulation problem of legs such as peripheral arterial occlusive disease or deep vein thrombosis;
3. had wounds or skin lesions over legs; and
4. had taken any medications which affect ANS activity.

Ages: 16 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Healthy female students aged 16-20 years with primary dysmenorrhea
Enrollment: 68 (Actual)
Dates: Start 2013-12-15 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Pain visual analog scale, pre-test | Before the intervention of menstruation day 1
  Pain visual analog scale was fulfilled as pain assessment before the intervention of menstruation day 1. The pain visual analog scale uses the 10 cm horizontal scale with verbal descriptors, the pain intensity could be graded from "no pain" (score of 0)" to "worst imaginable pain" (score of 10).
Pain visual analog scale, post-test | After the intervention of menstruation day 2
  Pain visual analog scale was fulfilled as pain assessment after the intervention of menstruation day 2. The pain visual analog scale uses the 10 cm horizontal scale with verbal descriptors, the pain intensity could be graded from "no pain" (score of 0)" to "worst imaginable pain" (score of 10).
Short-Form McGill Pain Questionnaire, pre-test | Before the intervention of menstruation day 1
  Short-Form McGill Pain Questionnaire was fulfilled as pain assessment before the intervention of menstruation day 1. It consists of 15 descriptors including 11 descriptors in the sensory subscale and four descriptors in the affective subscale. The pain intensity is scored from "none" (score 0) to "severe" (score 3) for each descriptor, summing the total pain rate index score of 0-45.
Short-Form McGill Pain Questionnaire, post-test | After the intervention of menstruation day 2
  Short-Form McGill Pain Questionnaire was fulfilled as pain assessment after the intervention of menstruation day 2. It consists of 15 descriptors including 11 descriptors in the sensory subscale and four descriptors in the affective subscale. The pain intensity is scored from "none" (score 0) to "severe" (score 3) for each descriptor, summing the total pain rate index score of 0-45.
Heart rate variability, pre-test of day 1 | Before the interventions on day 1
  Heart rate variability was measured before the interventions on day 1 to assess autonomic nervous function for all participants. Under a sampling rate of 512 Hz, signals from a lead I electrocardiogram were documented by an 8-bit analog-to-digital converter. Fast Fourier transformation was utilized to perform power spectral analysis, which quantified the power spectrum into the standard frequency-domain measurements, including LF (0.04-0.15 Hz), HF (0.15-0.40 Hz) and LF/HF ratio.
Heart rate variability, post-test of day 1 | After the interventions on day 1
  Heart rate variability was measured after the interventions on day 1 to assess autonomic nervous function for all participants. Under a sampling rate of 512 Hz, signals from a lead I electrocardiogram were documented by an 8-bit analog-to-digital converter. Fast Fourier transformation was utilized to perform power spectral analysis, which quantified the power spectrum into the standard frequency-domain measurements, including LF (0.04-0.15 Hz), HF (0.15-0.40 Hz) and LF/HF ratio.
Heart rate variability, pre-test of day 2 | Before the interventions on day 2
  Heart rate variability was measured before the interventions on day 2 to assess autonomic nervous function for all participants. Under a sampling rate of 512 Hz, signals from a lead I electrocardiogram were documented by an 8-bit analog-to-digital converter. Fast Fourier transformation was utilized to perform power spectral analysis, which quantified the power spectrum into the standard frequency-domain measurements, including LF (0.04-0.15 Hz), HF (0.15-0.40 Hz) and LF/HF ratio.
Heart rate variability, post-test of day 2 | After the interventions on day 2
  Heart rate variability was measured after the interventions on day 2 to assess autonomic nervous function for all participants. Under a sampling rate of 512 Hz, signals from a lead I electrocardiogram were documented by an 8-bit analog-to-digital converter. Fast Fourier transformation was utilized to perform power spectral analysis, which quantified the power spectrum into the standard frequency-domain measurements, including LF (0.04-0.15 Hz), HF (0.15-0.40 Hz) and LF/HF ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Wu Shih-Ju, Principal Investigator — Saint Mary's Hospital Luodong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu SJ, Kan WC, Shiao CC. Warm-water footbath improves dysmenorrhoea and heart rate variability in college students: a randomised controlled trial. J Obstet Gynaecol. 2022 Jul;42(5):1204-1210. doi: 10.1080/01443615.2021.1945007. Epub 2021 Sep 24. PMID 34560833